CLINICAL TRIAL: NCT04427111
Title: Therapeutic Efficiency Analyses of Mandibular Advancement Devices on Obstructive Sleep Apnea Using Polysomnography, Smartphone Sleep Applications, and Simple Pulse Oximeter
Brief Title: Therapeutic Efficiency of Mandibular Advancement Device Using Smartphone Sleep Applications and Pulse Oximeter
Status: Completed | Type: Observational
Sponsor: Bahadır EZMEK (Other)
Responsible Party: Sponsor-Investigator, Bahadır EZMEK, Assistant Professor, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Organization: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Other Study IDs: 2015-KAEK-84
Record Dates: First submitted 2020-06-04; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Obstructive Sleep Apnea
Keywords: Snoring; Obstructive sleep apnea; Mandibular advancement device; Pulse oximeter device; Smartphone sleep applications
MeSH Terms: conditions — Sleep Apnea, Obstructive; Snoring

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mild-moderate OSA patients for MAD treatment: Patients are classified as mild Obstructive Sleep Apnea (OSA) if they have between 5-15 Apnea-Hypopnea Index, moderate if they have between 15-30, and severe if they have >30, as measured by Polysomnography (Epstein LJ, Kristo D, Strollo PJ, et al. 2009). The principal treatment methodology for OSA patients is positive airway pressure. In patients with mild to moderate OSA, oral appliances such as mandibular advancement devices (MAD) is alternately indicated (Ramar K, Dort LC, Katz SG, et al. 2015) The American Academy of Dental Sleep Medicine (Ramar K, Dort LC, Katz SG, et al. 2015) recommended titratable-customized MADs for patient comfort and the ability to permit modifications in the amount of mandibular protrusion for treatment efficacy. However, Aarab et al (Aarab G, Lobbezoo F, Hamburger HL, Naeije M. 2010) demonstrated similar therapeutic efficiency of non-titratable-customized MADs in the treatment of OSA
  Interventions: Device: Non-titratable-customized mandibular advancement device

INTERVENTIONS:
Device: Non-titratable-customized mandibular advancement device — The most comfortable protruded mandibular position situated between 60-75% of MMPV was determined according to patient response with 6mm of the vertical interocclusal dimension between maxillary and mandibular central incisors and registered. The upper and lower acrylic resin splints were secured to each other in the posterior region with auto polymerizing acrylic resin and NTC-MADs were obtained. The patients were instructed to wear their non-titratable-customized mandibular advancement device every night.

SUMMARY:
An observational clinical trial in a single centre. The objective of this study was to determine the efficacy of mandibular advancement device (MAD) therapy on snoring intensity, frequency, and oxygen desaturation periods in mild-moderate obstructive sleep apnea (OSA) patients with snoring problems. Totally, 18 mild-moderate OSA patients (8 females and 10 males) with subjective snoring complaint were selected. Each patient's diagnostic polysomnographic analysis (PSG) was accepted as initial PSG values. Each patient was subjected simple pulse oximeter (SPO) and smartphone sleep application (SSA) at 3 different nights at home. Diagnostic mean values of oxygen desaturation index (obtained by using SPO), snoring intensity score (obtained by using SSA), and snoring percentage (obtained by using SSA) were recorded. Non-titratable-customized MAD with 60-75% of maximal mandibular protrusion were fabricated. The patients were instructed to wear their MAD every night. SPO and SSA measurement were repeated at the 1st, 4th, 12th, and 24th week of the treatment process. At the 24th week of treatment, The PSG were repeated and all PSG, SPO, and SSA values were compared with initial diagnostic values.

ELIGIBILITY:
Inclusion Criteria:

* mild-moderate OSA patients with subjective snoring complaints

Exclusion Criteria:

* Severe OSA
* Undergone previous surgical therapy for SS or OSA
* High-risk of cardiovascular, respiratory, neurological, or psychiatric disorders
* Inadequate dental anchor for MAD treatment
* Temporomandibular joint dysfunction
* Angle Class III maxillomandibular relation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mild-moderate obstructive sleep apnea patients were referred Department of Prosthodontics, Gülhane Faculty of Dentistry for oral appliance treatment
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2015-12-24 (Actual); Primary Completion 2017-12-24 (Actual); Study Completion 2017-12-24 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Apnea-Hypopnea Index (AHI) at 6 months | at baseline and in 6 months
  AHI was defined as total number of apnea or hypopnea events which lasts for at least ten seconds per hour during full nigth polysomnography (PSG) and accepted to be the main physiological sleep parameter in the present study. The AHI values were used for the evaluation of the severity of OSA and the MAD's treatment success in OSA patients

SECONDARY OUTCOMES:
Oxygen-desaturation index (ODI) | at baseline and in 6 months
  ODI was used to evaluate the desaturation fluctuations during full night PSG. ODI is defined as 3-4% decrease in oxygen saturation per hour.
Snoring index (SI) | at baseline and in 6 months
  SI was used to evaluate snoring events per hour during PSG
Simple pulse oximeter (SPO)/ODI | at baseline and 1, 4, 12, and 24 week of MAD treatment
  SPO/ODI was used to evaluate the desaturation fluctuations during sleep in-home environment by using simple pulse oximeter device
Smartphone sleep application (SSA)/snoring intensity score (SIS) | at baseline and 1, 4, 12, and 24 week of MAD treatment
  SSA/SIS was used to evaluate snoring intensity that was calculated by SSA during sleep in-home environment. No information exists about how to calibrate the SSA to calculate SIS
SSA/snoring percentage (SP) | at baseline and 1, 4, 12, and 24 week of MAD treatment
  SSA/SP was the ratio of total snoring time to total sleep time that was calculated by SSA during sleep in-home environment. No information exists about how to calibrate the SSA to calculate SP.

CONTACTS AND LOCATIONS:
Overall Officials: Bulent Piskin, Prof., Study Chair — Technology of Dental Prosthodontics, Kapadokya University, Turkey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ramar K, Dort LC, Katz SG, Lettieri CJ, Harrod CG, Thomas SM, Chervin RD. Clinical Practice Guideline for the Treatment of Obstructive Sleep Apnea and Snoring with Oral Appliance Therapy: An Update for 2015. J Clin Sleep Med. 2015 Jul 15;11(7):773-827. doi: 10.5664/jcsm.4858. PMID 26094920
- [Result] Aarab G, Lobbezoo F, Hamburger HL, Naeije M. Effects of an oral appliance with different mandibular protrusion positions at a constant vertical dimension on obstructive sleep apnea. Clin Oral Investig. 2010 Jun;14(3):339-45. doi: 10.1007/s00784-009-0298-9. Epub 2009 Jun 18. PMID 19536571
- [Result] Zhou J, Liu YH. A randomised titrated crossover study comparing two oral appliances in the treatment for mild to moderate obstructive sleep apnoea/hypopnoea syndrome. J Oral Rehabil. 2012 Dec;39(12):914-22. doi: 10.1111/joor.12006. Epub 2012 Sep 27. PMID 23016888
- [Result] Fiz JA, Jane R, Sola-Soler J, Abad J, Garcia MA, Morera J. Continuous analysis and monitoring of snores and their relationship to the apnea-hypopnea index. Laryngoscope. 2010 Apr;120(4):854-62. doi: 10.1002/lary.20815. PMID 20222022
- [Result] Umemoto G, Toyoshima H, Yamaguchi Y, Aoyagi N, Yoshimura C, Funakoshi K. Therapeutic Efficacy of Twin-Block and Fixed Oral Appliances in Patients with Obstructive Sleep Apnea Syndrome. J Prosthodont. 2019 Feb;28(2):e830-e836. doi: 10.1111/jopr.12619. Epub 2017 Apr 19. PMID 28422345
- [Result] Isacsson G, Fodor C, Sturebrand M. Obstructive sleep apnea treated with custom-made bibloc and monobloc oral appliances: a retrospective comparative study. Sleep Breath. 2017 Mar;21(1):93-100. doi: 10.1007/s11325-016-1377-1. Epub 2016 Jul 5. PMID 27380034
- [Result] Jobin V, Mayer P, Bellemare F. Predictive value of automated oxygen saturation analysis for the diagnosis and treatment of obstructive sleep apnoea in a home-based setting. Thorax. 2007 May;62(5):422-7. doi: 10.1136/thx.2006.061234. Epub 2007 Jan 24. PMID 17251319
- [Result] Ernst G, Bosio M, Salvado A, Dibur E, Nigro C, Borsini E. Difference between apnea-hypopnea index (AHI) and oxygen desaturation index (ODI): proportional increase associated with degree of obesity. Sleep Breath. 2016 Dec;20(4):1175-1183. doi: 10.1007/s11325-016-1330-3. Epub 2016 Mar 30. PMID 27026417
- [Result] Camacho M, Robertson M, Abdullatif J, Certal V, Kram YA, Ruoff CM, Brietzke SE, Capasso R. Smartphone apps for snoring. J Laryngol Otol. 2015 Oct;129(10):974-9. doi: 10.1017/S0022215115001978. Epub 2015 Sep 3. PMID 26333720
- [Result] Stippig A, Hubers U, Emerich M. Apps in sleep medicine. Sleep Breath. 2015 Mar;19(1):411-7. doi: 10.1007/s11325-014-1009-6. Epub 2014 Jun 3. PMID 24888483
- [Result] Walker-Engstrom ML, Ringqvist I, Vestling O, Wilhelmsson B, Tegelberg A. A prospective randomized study comparing two different degrees of mandibular advancement with a dental appliance in treatment of severe obstructive sleep apnea. Sleep Breath. 2003 Sep;7(3):119-30. doi: 10.1007/s11325-003-0119-3. PMID 14569523
- [Result] Lee CH, Mo JH, Choi IJ, Lee HJ, Seo BS, Kim DY, Yun PY, Yoon IY, Won Lee H, Kim JW. The mandibular advancement device and patient selection in the treatment of obstructive sleep apnea. Arch Otolaryngol Head Neck Surg. 2009 May;135(5):439-44. doi: 10.1001/archoto.2009.31. PMID 19451462
- [Result] Petri N, Svanholt P, Solow B, Wildschiodtz G, Winkel P. Mandibular advancement appliance for obstructive sleep apnoea: results of a randomised placebo controlled trial using parallel group design. J Sleep Res. 2008 Jun;17(2):221-9. doi: 10.1111/j.1365-2869.2008.00645.x. PMID 18482111
- [Result] Nerfeldt P, Friberg D. Effectiveness of Oral Appliances in Obstructive Sleep Apnea with Respiratory Arousals. J Clin Sleep Med. 2016 Aug 15;12(8):1159-65. doi: 10.5664/jcsm.6058. PMID 27397661